CLINICAL TRIAL: NCT00712907
Title: Effects of Vitamin C on Hyperoxia-Induced Reduction of Retinal Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjäger-Mayrl, MD, Department of Clinical Pharmacology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: OPHT-161202
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Ocular Physiology; Regional Blood Flow
Keywords: vitamin C; retinal blood flow; intraocular pressure; retinal vessel diameter
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): vitamin C (Mayrhofer)
  Interventions: Dietary Supplement: vitamin C (Mayrhofer) 24mg/min i.v. for 64 min; Other: 100% O2 (AGA) two times for 12 min
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo; Other: 100% O2 (AGA) two times for 12 min

INTERVENTIONS:
Dietary Supplement: vitamin C (Mayrhofer) 24mg/min i.v. for 64 min — Substance: Ascorbic acid (Mayrhofer) Manufacturer: Mayrhofer, Linz, Austria Dosage form: i.v. Dosage: 24mg/min over 64 min Dosage reference: Ting HH 1996
  Arms: 1
Dietary Supplement: Placebo — Substance: Physiologic saline solution 0.9% (placebo) Dosage form: i.v. Dosage: 24ml/min over 64 min
  Arms: 2
Other: 100% O2 (AGA) two times for 12 min — Substance: 100% oxygen (AGA, Vienna, Austria, gases for human use) Manufacturer: AGA, Vienna, Austria, gases for human use Dosage form: Inhalation through an oxygenmask over a period of 12 minutes two times per study day.
  Dosage reference: Strenn K 1997

SUMMARY:
High arterial blood oxygen tension leads to vasoconstriction of retinal vessels, possibly related to an interaction between reactive oxygen species and endothelium-derived vasoactive factors. Vitamin C is a potent antioxidant capable of reversing endothelial dysfunction due to increased oxidant stress. Vitamin C appears to have vasodilatory properties, but the underlying mechanisms are not well understood.

In the present study we hypothesized that hyperoxic vasoconstriction of retinal vessels could be diminished by vitamin C.

Ocular blood flow will be determined by non-invasive methods, including laser Doppler velocimetry and the Zeiss retinal vessel analyser.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must A 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2003-02; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Retinal arterial and venous diameter (Zeiss retinal vessel analyzer) | in total 6 hours
Retinal blood flow velocity (laser Doppler velocimetry) | in total 6 hours
Intraocular pressure (applanation tonometry) | in total 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria